CLINICAL TRIAL: NCT06849557
Title: Effectiveness of Chair-bound Exergaming on Physical and Cognitive Functions in Pre-frail/ Frail Older Adults in Nursing Home: A Pilot Randomized Controlled Trial
Brief Title: Chair-bound Exergaming in Pre-frail/ Frail Older Adults in Nursing Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HE-SF2024/58
Record Dates: First submitted 2025-01-16; First posted 2025-02-27 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-01

CONDITIONS: Frailty in Older Adults
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-list Control (No Intervention): Wait list control, after post-test, 12 week supervised exercise intervention
- Exergaming (Experimental): 12-week exergaming intervention
  Interventions: Behavioral: Exergaming

INTERVENTIONS:
Behavioral: Exergaming — This intervention will last 12 weeks. Frail/ pre-frail participants will engage in supervised chair-bound exergaming.
  Arms: Exergaming

SUMMARY:
This pilot randomized controlled trial is designed to investigate the effectiveness of chair-bound exergaming on improving physical and cognitive function in pre-frail/ frail nursing home residents

DETAILED DESCRIPTION:
Objective To explore the effects of the chair-bound exergaming on the enjoyment of physical activity in in pre-frail/ frail nursing home residents.

To evaluate the effects of the chair-bound exergaming in improving physical and cognitive function in pre-frail/ frail nursing home residents.

Research plan and methodology Thirty nursing home residents will be recruited from the nursing homes.

All the eligible participant will be randomly allocated to either one of the following 2 groups (i) Exergaming (intervention group), or (ii) wait list control.

1. Intervention group (exergaming group, ERG) Those allocated to the ERG will receive supervised chair-bound exercise programme for 12 weeks.
2. Control group (wait list control, CG) Those allocated to the CG will receive supervised chair-bound exercise programme for 12 weeks after post-assessment.

ELIGIBILITY:
Inclusion Criteria:

* older adults aged 60 years or older living in the nursing homes;
* pre-frail or frail according to the Fried Frailty Phenotypes;
* ability to understand and execute instructions; and
* ability to sit unassisted on a chair or in a wheelchair.

Exclusion Criteria:

* no controlled medical diagnosed of severe cardiometabolic, respiratory and musculoskeletal disorders;
* any conditions that hinder the participation of intervention and assessment; and
* being involved in any other clinical trials.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
upper extremity endurance | T0: baseline
  upper extremity endurance measured by arm curl test
upper extremity endurance | T1: 6 week
  upper extremity endurance measured by arm curl test
upper extremity endurance | T2: immediately (1 week) after intervention
  upper extremity endurance measured by arm curl test
enjoyment | T0: baseline
  enjoyment of physical activity measured by Physical Activity Enjoyment Scale (PACES)
enjoyment | T1: 6 week
  enjoyment of physical activity measured by Physical Activity Enjoyment Scale (PACES)
enjoyment | T2: immediately (1 week) after intervention
  enjoyment of physical activity measured by Physical Activity Enjoyment Scale (PACES)

SECONDARY OUTCOMES:
upper extremity strength | T0: baseline
  upper extremity strength measured by handheld dynamometer
upper extremity strength | T1: 6 week
  upper extremity strength measured by handheld dynamometer
upper extremity strength | T2: immediately (1 week) after intervention
  upper extremity strength measured by handheld dynamometer
lung capacity | T0: baseline
  lung capacity measured by peak flow meter
lung capacity | T1: 6 week
  lung capacity measured by peak flow meter
lung capacity | T2: immediately (1 week) after intervention
  lung capacity measured by peak flow meter
sitting balance | T0: baseline
  sitting balance measured by sitting with opened eyes, sitting with closed eyes, sitting with shaking "no" and sitting with lifted leg
sitting balance | T1: 6 week
  sitting balance measured by sitting with opened eyes, sitting with closed eyes, sitting with shaking "no" and sitting with lifted leg
sitting balance | T2: immediately (1 week) after intervention
  sitting balance measured by sitting with opened eyes, sitting with closed eyes, sitting with shaking "no" and sitting with lifted leg
feasibility, acceptability and appropriateness of intervention | T2: immediately (1 week) after intervention
  feasibility, acceptability and appropriateness of intervention measured by questionnaire
mental health | T0: baseline
  mental health measured by Patient Health Questionnaire-4 (PHQ-4), range: 0-12; higher score indicates more psychological distress
mental health | T1: 6 week
  mental health measured by Patient Health Questionnaire-4 (PHQ-4), range: 0-12; higher score indicates more psychological distress
mental health | T2: immediately (1 week) after intervention
  mental health measured by Patient Health Questionnaire-4 (PHQ-4), range: 0-12; higher score indicates more psychological distress
cognitive function | T0: baseline
  cognitive function measured by Montreal Cognitive Assessment (MoCA), range: 0-30; lower score indicates more cognitive impairment.
cognitive function | T1: 6 week
  cognitive function measured by Montreal Cognitive Assessment (MoCA), range: 0-30; lower score indicates more cognitive impairment.
cognitive function | T2: immediately (1 week) after intervention
  cognitive function measured by Montreal Cognitive Assessment (MoCA), range: 0-30; lower score indicates more cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hiu Kwong (Tak Yue) Nursing Centre, Kowloon, Hong Kong